CLINICAL TRIAL: NCT02046850
Title: A Phase I Open-label, Single-center Study to Assess the Effect of the CYP3A4 Inducer Rifampicin on the Pharmacokinetics of a 75 mg Single Oral Dose of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Healthy Volunteers Aged 18 to 45 Years
Brief Title: To Assess the Effect of Rifampicin on the Pharmacokinetics of Selumetinib in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: D1532C00085
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2014-04-29 (Estimated); Status verified 2014-04

CONDITIONS: Solid Tumours
Keywords: Phase I, healthy, pharmacokinetics,
MeSH Terms: interventions — AZD 6244; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- selumetinib 75mg. (Experimental): Volunteers will receive selumetinib 75mg administered by mouth, as a capsule
  Interventions: Drug: selumetinib
- rifampicin 600mg. (Other): Volunteers will receive rifampicin 600mg administered by mouth, as a capsule
  Interventions: Drug: rifampicin
- selumetinib 75mg and rifampicin 600mg (Experimental): Volunteers will receive selumetinib 75mg and rifampicin 600mg, by mouth, as a capsule
  Interventions: Drug: selumetinib; Drug: rifampicin

INTERVENTIONS:
Drug: selumetinib — Volunteers will receive a single oral dose of 75 mg selumetinib on day 1 (Treatment A).
  Other Names: AZD6244
  Arms: selumetinib 75mg.
Drug: rifampicin — Volunteers will receive single, daily, oral doses of 600 mg rifampicin on Days 4 to 11 (Treatment B).
  Other Names: AZD6244
  Arms: rifampicin 600mg.
Drug: selumetinib — On day 12 volunteers will receive a single oral dose of 75 mg selumetinib (Treatment C).
  Arms: selumetinib 75mg and rifampicin 600mg
Drug: rifampicin — On day 12 volunteers will receive a single oral dose of 600 mg rifampicin. Once daily rifampicin administrations will continue through to Day 14 (Treatment C).
  Arms: selumetinib 75mg and rifampicin 600mg

SUMMARY:
Study to assess the effect of Rifampicin on the pharmacokinetics of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Healthy Male Volunteers

DETAILED DESCRIPTION:
A Open-label, Single-center Study to Assess the Effect of the CYP3A4 inducer Rifampicin on the Pharmacokinetics of a 75 mg Single Oral Dose of Selumetinib (AZD6244; ARRY-142886) (Hyd-Sulfate) in Healthy Volunteers

ELIGIBILITY:
Inclusion Criteria: 1. Have a body mass index (BMI) between 18 and 30 kg/m2 (inclusive) and weigh at least 50 kg and no more than 100 kg (inclusive). 2. Must not have smoked or used nicotine products within the previous 3 months. 3. Have a calculated creatinine clearance (CrCL) greater than 50 mL/min using the Cockcroft-Gault formula.

Exclusion Criteria: 1. Subjects of Japanese or non-Japanese Asian ethnicity. 2. Any one parent or grandparent (maternal or paternal) is Japanese or non-Japanese Asian (eg, China, Taiwan, Korea, Philippines, Thailand, Vietnam and Malaysia). Asian Indians are acceptable. 3. Current or past history of central serous retinopathy or retinal vein thrombosis,intra-ocular pressure greater than 21 mmHg or uncontrolled glaucoma. 4. Any clinically relevant abnormal findings in physical examination, hematology, clinical chemistry, urinalysis, vital signs or ECG at baseline in the opinion of the investigator. 5. History of presence of any clinically significant disease or disorder in the opinion of the investigator.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2014-02; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of selumetinib by assessment of area under the plasma concentration-time curve from time zero to infinity (AUC) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments

SECONDARY OUTCOMES:
Pharmacokinetics of selumetinib, N-desmethyl selumetinib,(and the amide metabolite, if deemed appropriate) by assessment of area under the plasma concentration-time from time zero to the time of the last quantifiable concentration (AUC(0-t) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, N-desmethyl selumetinib,(and the amide metabolite, if deemed appropriate) by assessment of area under the plasma concentration-time curve from time zero to 12 hours post-dose AUC(0-12) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, N-desmethyl selumetinib,(and the amide metabolite, if deemed appropriate) by assessment of maximum plasma concentration (Cmax) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, N-desmethyl selumetinib,(and the amide metabolite, if deemed appropriate) by assessment of time to Cmax (tmax) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, by assessment of apparent systemic plasma clearance (CL/F) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, by assessment of apparent volume at distribution equilibrium, mean residence time (MRT)*CL/F (Vss/F) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, by assessment of apparent volume at distribution (Vz/F) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, N-desmethyl selumetinib,(and the amide metabolite, if deemed appropriate) by assessment of terminal half-life (t1/2) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib, N-desmethyl selumetinib,(and the amide metabolite, if deemed appropriate) by assessment of terminal rate constant (λz) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assessment of AUC metabolite to parent ratio, n-desmethyl selumetinib (MRAUC) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib and N-desmethyl selumetinib by assessment of Cmax metabolite to parent ratio, n-desmethyl selumetinib (MRCmax) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments
Pharmacokinetics of selumetinib by assessment of mean residence time (MRT) | Blood samples are collected pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 24, 36, 48 and 72 hours post dose
  Samples taken during each of the 3 treatments

OTHER OUTCOMES:
Safety variables (adverse events, physical examinations, ophthalmologic assessments, vital signs, clinical laboratory assessments, and 12 lead electrocardiograms) | Baseline (Day-1) up to Day 25
  Assessments performed during each of the 3 treatments

CONTACTS AND LOCATIONS:
Overall Officials: Eleanor Lisbon, MD, Principal Investigator — Quintiles 6700 W 115th Street, Kansas, US
Locations (1):
- Research Site, Overland Park, Kansas, United States